CLINICAL TRIAL: NCT05525793
Title: Effectiveness of the Transitional Care Model in Total Knee Arthroplasty Patients: A Randomized Controlled Study
Brief Title: Effectiveness of the Transitional Care Model in Total Knee Arthroplasty Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Ayla Güllü, Principal Investigator, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Hasan Kalyoncu Üniversitesi; 2021/004 (Other: Scientific Research Ethical Board)
Record Dates: First submitted 2022-08-25; First posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Knee Osteoarthritis; Pain; Self Efficacy; Health Care Utilization
MeSH Terms: conditions — Osteoarthritis, Knee; Pain; Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transitional care (Experimental): This group is the actual intervention group.
  Interventions: Other: Transitional care model
- Usual care (No Intervention): This group is the routine treatment (control) valid in the clinical practice.

INTERVENTIONS:
Other: Transitional care model — The patients who were assigned to this group with the transitional care model, 6 weeks of counseling and intervention training provided continuity of care and a safe transition, and patients were encouraged about symptom management and a healthy lifestyle.
  Arms: Transitional care

SUMMARY:
The aim of this study was to determine the effectiveness of transitional care in patients with total knee arthroplasty on patients' functional status, perceived self-efficacy, and health care use. Based on the sampling inclusion criteria, we assigned the patients who would undergo knee arthroplasty to the control (n=35) and intervention (n=35) groups, via the block randomization method. The intervention group received transitional care, while the control group received usual care. Data were collected on post-intervention functional status, level of self-efficacy, and hospital visits outside of routine control.

DETAILED DESCRIPTION:
This randomised control study was conducted 70 eligible partients with total knee arthroplasty in a public hospital orthopedic and traumatology service. Participants were randomly assigned to receive either the 6-week 'Transitional Care Model' program or usual care. Assessments of self-efficacy and functional status of patients were conducted at baseline, 2nd and 9th weeks after discharge. Time-dependent changes in patient outcomes were assessed by using Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and Arthritis Self-efficacy Scale (ASES) measurements tools. Assessments of hospital visits outside of routine control were conducted 2nd week, 6th week, 9th week, and 12th weeks after discharge. The functional status of the intervention group patients improved more than the control group according to WOMAC mean scores. Intervention group patients receiving transitional care had higher mean scores at the 2nd-week and 9th-week postoperatively in perceived self-efficacy . Besides, the rate of admission to the hospital in the intervention group was lower compared to the control group, and a significant difference was observed in the 6th-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Having decided to undergo total knee arthroplasty for the first time due to osteoarthritis
* Volunteering to participate in the research, not having a psychological, physical, and mental disability that may prevent communication, not having any major chronic problems such as end-stage organ failure, kidney, neurological, cancer
* Being discharged to the home from a hospital
* Being able to speak Turkish
* Being available by phone
* Being aged 50 and over

Exclusion Criteria:

* Unwillingness to continue the study
* Rehospitalization
* Exposure to a disease or trauma that would affect functional independence during the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-08-08 (Actual); Study Completion 2021-11-11 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index-WOMAC | up to 9 weeks
  Assessments of functional status of patients were conducted at baseline, 2nd and 9th weeks after discharge.
Arthritis Self-efficacy Scale (ASES) | up to 9 weeks
  Assessments of self-efficacy of patients were conducted at baseline, 2nd and 9th weeks after discharge.

SECONDARY OUTCOMES:
number of hospital visits | up to 12 weeks
  Assessments of the number of hospital visits outside of routine control were conducted 2nd week, 6th week, 9th week, and 12th weeks after discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Betül Tosun, Assoc. Prof., Study Chair — Hasan Kalyoncu Üniversitesi
Locations (1):
- Mustafa Kemal Üniversitesi, Antakya, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] An S, Li J, Xie W, Yin N, Li Y, Hu Y. Extracorporeal shockwave treatment in knee osteoarthritis: therapeutic effects and possible mechanism. Biosci Rep. 2020 Nov 27;40(11):BSR20200926. doi: 10.1042/BSR20200926. PMID 33074309
- [Background] Gaffney CJ, Pelt CE, Gililland JM, Peters CL. Perioperative Pain Management in Hip and Knee Arthroplasty. Orthop Clin North Am. 2017 Oct;48(4):407-419. doi: 10.1016/j.ocl.2017.05.001. Epub 2017 Jun 29. PMID 28870302
- [Background] Magan AA, Ahmed SS, Paton B, Konan S, Haddad FS. Does Multimodal Therapy Influence Functional Outcome After Total Knee Arthroplasty? Orthop Clin North Am. 2020 Oct;51(4):453-459. doi: 10.1016/j.ocl.2020.06.011. PMID 32950214
- [Background] Hanusch BC, O'Connor DB, Ions P, Scott A, Gregg PJ. Effects of psychological distress and perceptions of illness on recovery from total knee replacement. Bone Joint J. 2014 Feb;96-B(2):210-6. doi: 10.1302/0301-620X.96B2.31136. PMID 24493186
- [Background] Mardani A, Griffiths P, Vaismoradi M. The Role of the Nurse in the Management of Medicines During Transitional Care: A Systematic Review. J Multidiscip Healthc. 2020 Oct 30;13:1347-1361. doi: 10.2147/JMDH.S276061. eCollection 2020. PMID 33154651
- [Background] Allen J, Hutchinson AM, Brown R, Livingston PM. Communication and Coordination Processes Supporting Integrated Transitional Care: Australian Healthcare Practitioners' Perspectives. Int J Integr Care. 2020 Apr 16;20(2):1. doi: 10.5334/ijic.4685. PMID 32322183
- [Result] Morkisch N, Upegui-Arango LD, Cardona MI, van den Heuvel D, Rimmele M, Sieber CC, Freiberger E. Components of the transitional care model (TCM) to reduce readmission in geriatric patients: a systematic review. BMC Geriatr. 2020 Sep 11;20(1):345. doi: 10.1186/s12877-020-01747-w. PMID 32917145
- [Result] Hung D, Leidig RC. Implementing a transitional care program to reduce hospital readmissions among older adults. J Nurs Care Qual. 2015 Apr-Jun;30(2):121-9. doi: 10.1097/NCQ.0000000000000091. PMID 25485791
- [Result] Costa MFBNAD, Sichieri K, Poveda VB, Baptista CMC, Aguado PC. Transitional care from hospital to home for older people: implementation of best practices. Rev Bras Enferm. 2020 Nov 2;73Suppl 3(Suppl 3):e20200187. doi: 10.1590/0034-7167-2020-0187. eCollection 2020. English, Portuguese. PMID 33146267
- [Result] Lyu QY, Huang JW, Li YX, Chen QL, Yu XX, Wang JL, Yang QH. Effects of a nurse led web-based transitional care program on the glycemic control and quality of life post hospital discharge in patients with type 2 diabetes: A randomized controlled trial. Int J Nurs Stud. 2021 Jul;119:103929. doi: 10.1016/j.ijnurstu.2021.103929. Epub 2021 Mar 26. PMID 33901941
- [Result] Liu ZC, Gao L, Zhang WH, Wang J, Liu RR, Cao BH. Effects of a 4-week Omaha System transitional care programme on rheumatoid arthritis patients' self-efficacy, health status, and readmission in mainland China: A randomized controlled trial. Int J Nurs Pract. 2020 Aug;26(4):e12817. doi: 10.1111/ijn.12817. Epub 2020 Jan 27. PMID 31985129
- [Result] Kranker K, Barterian LM, Sarwar R, Peterson GG, Gilman B, Blue L, Stewart KA, Hoag SD, Day TJ, Moreno L. Rural hospital transitional care program reduces Medicare spending. Am J Manag Care. 2018 May;24(5):256-260. PMID 29851443
- [Result] Nall RW, Herndon BB, Mramba LK, Vogel-Anderson K, Hagen MG. An Interprofessional Primary Care-Based Transition of Care Clinic to Reduce Hospital Readmission. Am J Med. 2020 Jun;133(6):e260-e268. doi: 10.1016/j.amjmed.2019.10.040. Epub 2019 Dec 24. PMID 31877267